CLINICAL TRIAL: NCT03029013
Title: A Phase II Clinical Trial Study on Apatinib and Chemotherapy Sequential Treatment With Advanced Metastatic Cervical Cancer
Brief Title: Apatinib and Chemotherapy Sequential Treatment With Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ge Wang, M.D., Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACSTCC
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — apatinib

ARMS (1):
- experimental group (Experimental): Apatinib and chemotherapy
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib， 250 mg qd，po，after 7 days , paclitaxel (135-175 mg/m2) and platinum two drug standard chemotherapy, 21 days as a treatment cycle，during the chemotherapy of 7-21 days continue to offer the Apatinib. without disease progress, after 4 chemotherapy cycles, patients continue to accept the Apatinib maintenance treatment.
  Other Names: YN968D1

SUMMARY:
The study is the single arm and single center clinical trials，We conduct the phase II clinical trial to further explore the efficacy and safety of Apatinib and chemotherapy sequential treatment with advanced recurrence of metastatic cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis of recurrent or metastatic cervical cancer;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1;
* Life expectancy of more than 3months;
* With normal marrow, liver and renal function：

  * blood routine examination ：HB≥90g/L，ANC ≥1.5×10*9/L，PLT≥80×10*9/L；
  * Biochemical examination: total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL)，alanine aminotransferase (ALT) and aspartate aminotransferase (AST) of ≤2.5 UNL or ≤5 UNL ，acreatinine (Cr) of ≤ 1.25 UNL; creatinine clearance rate ≥ 45ml/min (Cockcroft-Gault);
* With written informed consent signed voluntarily by patients themselves .
* With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

* Uncontrolled hypertension
* Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias
* With abnormal coagulation function， bleeding tendency or treating with thrombolysis and anticoagulation
* History of clinically relevant major bleeding event (e.g. gastrointestinal hemorrhage, bleeding ulcer, occult blood ≥ (++), and vasculitis) =< 3 months prior to randomization;
* uncured the wound or fracture
* Centrally located tumors of local invasion of major blood vessels, or Researchers think that patients may invade the important blood vessels and cause fatal bleeding (CT or MRI);
* Factors affecting the oral medication (e.g. inability to swallow, chronic diarrhea and intestinal obstruction);
* Urine protein >++, or urine protein in 24 hours> 1.0g
* Accumulation of coelomic fluid (e.g. pleural effusion, ascites fluid, cardiac effusion) requiring treatment
* History of uncontrolled psychotropic drug abuse or mental disorders;
* Prior VEGFR inhibitor treatment ;
* Other malignancy within Before or at the same time other than basal cell skin cancer, or carcinoma in situ of the cervix;

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months

SECONDARY OUTCOMES:
overall survival | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China